CLINICAL TRIAL: NCT06167083
Title: Machine Learning in the ICU: Predicting Mortality in Patients With Carbapenem-Resistant Gram-Negative Bacilli Bloodstream Infections
Brief Title: Machine Learning in the ICU: Predicting Mortality in Bloodstream Infections (ICU:Intensive Care Unit)
Acronym: ICU
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Özlem Güler, Phd Medical Doctor, Kocaeli University
Other Study IDs: GOKAEK-2023/12.31
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Carbapenem Resistant Bacterial Infection
Keywords: Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deceased Patients: Carbapenem-resistant Gram-negative bacilli Blood Stream Infection With mortality
  Interventions: Diagnostic Test: Machine Learning to Estimate Mortality
- Surviving Patients: Carbapenem-resistant Gram-negative bacilli Blood Stream Infection Without mortality
  Interventions: Diagnostic Test: Machine Learning to Estimate Mortality

INTERVENTIONS:
Diagnostic Test: Machine Learning to Estimate Mortality — Using deep learning we try to develop an algorithm and anticipate mortality

SUMMARY:
Using our own patient data, our study aimed to predict mortality that can develop in Carbapenem-resistant Gram-negative bacilli bloodstream infections with a machine learning-based model.

In the intensive care unit, patients with bloodstream infections, both with and without mortality, will be examined retrospectively in two subgroups for comparison.

DETAILED DESCRIPTION:
Carbapenems are one of the last-resort antibiotics used to treat severe infections caused by multi-drug resistant Gram-negative pathogens. Infections with Carbapenem-resistant Gram-negative bacilli (CR-GNB) have become widespread in the past decade, posing serious threats to public health. Carbapenem-resistant Enterobacteriaceae (CRE), Carbapenem-resistant Acinetobacter baumannii (CRAB), and Carbapenem-resistant Pseudomonas aeruginosa (CRPA) top the priority list of antibiotic-resistant bacteria worldwide. CR-GNB causes a broad spectrum of infections, including bacteremia, urinary tract infections, pneumonia, and intra-abdominal infections. Carbapenem-resistant bloodstream infections are a significant cause of morbidity and mortality, and therapeutic options in treatment are extremely limited. By evaluating risk factors in patients monitored in the intensive care unit, scoring systems that can predict prognosis reduce mortality risk by ensuring the early application of effective antibiotics and timely hemodynamic support that are currently in use.

With the accumulation of big data and advancements in data storage techniques, innovative and pragmatic machine learning methods that have entered our lives demonstrate good prediction performance in the medical field. Machine learning-based models developed to predict mortality in patients monitored in the intensive care unit are available in the literature and provide an opportunity for earlier intervention in patients.

Using our own patient data, In the intensive care unit, patients with bloodstream infections, both with and without mortality, will be examined retrospectively in two subgroups for comparison. The investigators aim to predict mortality that can develop in Carbapenem-resistant Gram-negative bacilli bloodstream infections with a machine learning-based model.

ELIGIBILITY:
Inclusion Criteria:

* In our study, patients who were monitored in our hospital's tertiary Intensive Care Unit between June 2017 and June 2023 and developed bloodstream infections with Carbapenem-resistant Enterobacteriaceae, Carbapenem-resistant Acinetobacter baumannii and Carbapenem-resistant Pseudomonas aeruginosa will be retrospectively included.

Exclusion Criteria:

* Patients under the age of 18 and those with infections other than bloodstream infections will not be included.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who were monitored in our tertiary intensive care unit for six years retrospectively and developed bloodstream infections with Carbapenem-resistant Enterobacteriaceae, Acinetobacter baumannii and Pseudomonas aeruginosa have been included in the study with their personal data anonymized
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Risk of Mortality | 3 months
  The sensitivity and specificity will be defined with AUC-ROC curve (Area Under the Receiver Operating Characteristic curve) using machine learning algorithm

CONTACTS AND LOCATIONS:
Overall Officials: özlem güler, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Using machine learning methods to predict in-hospital mortality of sepsis patients in the ICU — https://bmcmedinformdecismak.biomedcentral.com/articles/10.1186/s12911-020-01271-2